CLINICAL TRIAL: NCT05832359
Title: Evaluation of Dental Maturation and Mandibular Bone Morphology in Childhood Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MUDHFP10
Record Dates: First submitted 2022-12-14; First posted 2023-04-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Childhood Rheumatic Diseases
Keywords: Childhood rheumatic diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children diagnosed with childhood rheumatic disease (Experimental)
  Interventions: Radiation: Panoramic rad.
- Healthy children (Experimental)
  Interventions: Radiation: Panoramic rad.

INTERVENTIONS:
Radiation: Panoramic rad. — In the study, digital panoramic x-rays of the patients will be evaluated and dental age estimation with Willems method and mandibular bone morphometric measurements will be made.

SUMMARY:
The aim of our study is to examine possible disease-related changes in dental age and mandibular bone morphology in childhood rheumatic diseases.

DETAILED DESCRIPTION:
to reveal the changes that can occur in different childhood rheumatic diseases, the treatment process of the disease and the drugs used on the dental age and mandible

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 14 years with childhood rheumatism
* Patients without bilateral congenital germ deficiency in the lower teeth
* Patients with seven teeth (except no #8) on the left of the mandibula (No seven teeth on the left of the mandibula, there should be a symmetrical tooth on the right of the mandibula.

Exclusion Criteria:

* Patients with bilateral congenital germ deficiency in lower teeth in intraoral and/or radiographic examinations
* Patients with asymmetry and magnification errors and where anatomical structures cannot be seen clearly in the panoramic x-ray
* Patients with a significant number of missing teeth due to trauma or disease, root canal treatment, and pathological tooth structure
* Patients with a history of other chronic diseases

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female/Male
Enrollment: 278 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Dental Age Estimation | 3 months
  The study group will be comprised of newly diagnosed pediatric patients who applied to Umraniye Training and Research Hospital Division of Pediatric Rheumatology and whose treatment is ongoing, and the control group will be composed of pediatric patients without systemic disease who applied to Marmara University Faculty of Dentistry Department of Pedodontics. In the study, digital panoramic x-rays of the patients will be evaluated and dental age estimation with Willems method will be made.

SECONDARY OUTCOMES:
Mandibular bone morphometric measurements | 3 months
  The study group will be comprised of newly diagnosed pediatric patients who applied to Umraniye Training and Research Hospital Division of Pediatric Rheumatology and whose treatment is ongoing, and the control group will be composed of pediatric patients without systemic disease who applied to Marmara University Faculty of Dentistry Department of Pedodontics.For mandibular bone morphometric measurements, fractal analysis, that is a mathematical method describing and analyzing complex shapes and structural patterns such as the bone tissue, will be used in order to assess the bone density, using Image J software. A region of interest will be selected from panoramic radiographs. Image processing will be applied to correct for lightning irregularity, and box-counting method will be used to calculate a fractal dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Ecem Ipek, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No